CLINICAL TRIAL: NCT04680091
Title: A Single-Center, Single-Arm, Open-Label, Fixed-Sequence Phase I Drug-Drug Interaction Clinical Study of the Effect of Efavirenz on Pharmacokinetics of Maleate Pyrotinib in Chinese Healthy Subjects.
Brief Title: Drug-Drug Interaction of Pyrotinib With a Moderate CYP3A Inducer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-DDI-05
Record Dates: First submitted 2020-10-21; First posted 2020-12-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2020-10

CONDITIONS: Healthy Subjects, Drug-drug Interaction, Pyrotinib
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Intervention Model Description: To observe the effect of efavirenz on the pharmacokinetics of pyrotinib and to evaluate the safety of pyrotinib, efavirenz and their coadministration in Chinese healthy subjects. The subjects will take pyrotinib at first single dose, then washout period, and take it at second single dose after multiple administration of efavirenz to get a full induction condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efavirenz 600 mg + Pyrotinib 400 mg (Experimental)
  Interventions: Drug: Pyrotinib Maleate; Drug: Efavirenz
- Pyrotinib 400 mg (Active Comparator)
  Interventions: Drug: Pyrotinib Maleate

INTERVENTIONS:
Drug: Pyrotinib Maleate — single oral dose, 400 mg, fed.
Drug: Efavirenz — single oral dose, 600 mg, fasted, at bedtime.
  Arms: Efavirenz 600 mg + Pyrotinib 400 mg

SUMMARY:
This drug-drug interaction (DDI) study had been designed to investigate the effect of a moderate CYP 3A inducer efavirenz on the pharmacokinetics of maleate pyrotinib in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
* Ability to complete the study as required by the protocol;
* Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
* Body weight ≥ 50 kg for male and female, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);
* In females, documented surgical sterilization, postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum at Screening), or agreement to use an approved form of contraception
* In males, agreement to avoid sperm donation for 6 months days after the dose of pyrotinib
* Liver function test results must be below the upper limit of normal.
* Participants must agree to refrain from donation of whole blood and other blood products from 90 days prior to Screening,

Exclusion Criteria:

* Loss of more than 400 mL blood during the 3 months before the trial (eg, as a blood donor)
* Allergic constitution;
* History of drug use, or drug abuse screening positive;
* Alcoholic or often drinkers;
* A smoker with 5 cigarettes per day for more than 90 days;
* Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy participants), anti-treponema pallidum virus (TP), or antihuman immunodeficiency virus (HIV) Type 1 and Type 2 (all subjects)
* Use of any drugs or substances known to be inhibitors or inducers of CYP3A4/5 within 90 days from the first dose or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to pyrotinib administration and during the study.
* A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
* Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Summary of Pharmacokinetic parameters Maximum Plasma Concentration (Cmax) for pyrotinib. | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
Summary of Pharmacokinetic parameters Area Under the Plasma Concentration-time Curve from 0 to any time before the last quantifiable concentration (AUC0-t) for pyrotinib. | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
Summary of Pharmacokinetic parameters Area Under the Plasma Concentration-time Curve from 0 to infinite time (AUCinf) for pyrotinib. | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20

SECONDARY OUTCOMES:
Pharmacokinetics parameters (Tmax) of pyrotinib; | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
Pharmacokinetics parameters (T1/2) of pyrotinib; | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
Pharmacokinetics parameters (CL) of pyrotinib; | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
Pharmacokinetics parameters (Vd) of pyrotinib; | predose, 1, 2, 3, 4, 4.5, 5, 5.5, 7, 9, 12, 24, 48, 72, 96 h for Day1 and predose, 0.5, 1, 1.75, 2.5, 3.25, 4, 4.75, 5.5, 6.5, 8, 12, 24, 48, 72 h for Day20
The incidence and severity of adverse events/serious adverse events (based on NCI-CTCAE 5.0): Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination, vital signs, etc. | Baseline up to 14 days post last dose, up to approximately 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu HengRui Medicine Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No